CLINICAL TRIAL: NCT04226235
Title: Acute Effects of Yoga on Arterial Stiffness, Wave Reflection, and Blood Markers in Normotensive and Hypertensive Adults
Brief Title: Acute Effects of Vinyasa Yoga on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 530
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1-hour vinyasa yoga session (Experimental): One hour of vinyasa yoga was completed by all participants while following a DVD.
  Interventions: Behavioral: Yoga session

INTERVENTIONS:
Behavioral: Yoga session — a 1-hour yoga session was completed by all participants following a DVD.

SUMMARY:
The purpose of this investigation was to determine the acute effects of vinyasa yoga on arterial stiffness, wave reflection, and blood markers in normo- and hyper-tensive adults. To address this aim, fifteen normotensive adults and 15 adults with elevated blood pressure or stage 1 hypertension with a minimum of 3 months of yoga practice experience were enrolled. Carotid-femoral pulse wave velocity (cf-PWV), augmentation index (AIx), lipid profile, and glucose concentrations were assessed at baseline and immediately following a 1-hour vinyasa yoga session.

ELIGIBILITY:
Inclusion Criteria:

* Having normal (systolic blood pressure <120 mm Hg with a diastolic <80 mm Hg) or elevated blood pressure (systolic blood pressure 120-129 mm Hg) or stage 1 hypertension (systolic blood pressure 130-139 mm Hg or a diastolic blood pressure 80-89 mm Hg).
* Must have had at least 3 months of prior yoga experience.

Exclusion Criteria:

* A history of cardiovascular disease or cardiac events, pregnancy, infection within the last 4 weeks, chronic obstructive pulmonary disease (COPD), endocrine or renal disease, metabolic disorders, or debilitating muscular, joint and bone injury.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Arterial stiffness | Once before the yoga session
  Carotid-femoral pulse wave velocity
Arterial stiffness | Once immediately after the 1-hour yoga session
  Carotid-femoral pulse wave velocity
Wave reflection | Once before the yoga session
  Augmentation index
Wave reflection | Once immediately after the 1-hour yoga session
  Augmentation index

SECONDARY OUTCOMES:
Lipid profile | Once before the yoga session
  Blood samples obtained via finger stick and analyzed for total-, LDL-, and HDL-cholesterol and triglyceride concentrations using reflectance photometry.
Lipid profile | Once immediately after the 1-hour yoga session
  Blood samples obtained via finger stick and analyzed for total-, LDL-, and HDL-cholesterol and triglyceride concentrations using reflectance photometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas State University, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: No